CLINICAL TRIAL: NCT03574467
Title: Functional Outcomes of The Bobath Neurodevelopmental Treatment Approach Applied to Patients With Brain Tumors: Comparison With Stroke Patients
Brief Title: Functional Outcomes of The Bobath Approach on Patients With Brain Tumors: Comparison With Stroke Patients
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ceyhun Turkmen, Research Assistant, Hacettepe University
Other Study IDs: GO 18/25-13
Record Dates: First submitted 2018-06-11; First posted 2018-07-02 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Brain Neoplasms; Stroke, Acute
Keywords: brain neoplasms; stroke; rehabilitation
MeSH Terms: conditions — Brain Neoplasms; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bobath Approach Applied to Patient with Brain Tumors
  Interventions: Behavioral: Bobath Neurodevelopmental Treatment Approach
- Bobath Approach Applied to Patient with Stroke
  Interventions: Behavioral: Bobath Neurodevelopmental Treatment Approach

INTERVENTIONS:
Behavioral: Bobath Neurodevelopmental Treatment Approach — The Bobath Neurodevelopmental Treatment (NDT) rehabilitation approach is effective in increasing the functional capacity and acquiring independence in patients with stroke and brain tumor.

SUMMARY:
The aim of this study is to examine the functional recovery results of the Bobath (NDT) approach in patients with primary brain tumors and compare the results with those of stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* acute phase patients with brain tumor and stroke in after surgery

Exclusion Criteria:

* Modified rankin scale <2
* High grade tumor
* Infratentorial tumor
* GCS<14
* Rehabilitation session time<3
* Second or more tumor surgery
* Second or more stroke
* Bilateral stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Department of Neurology between June 2016 and April 2017, were analyzed for the study. The study inclusion criteria were determined for all patients to be over 18 years of age, in the acute phase, Glasgow Coma Scale score 14 and above, Modifiye Rankin Score being more than 2 and medical stability. Furthermore, the criteria for inclusion in the study were unilateral stroke and having a stroke for the first time for stroke patients, and supratentorial location for patients with brain tumors.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-06-12 (Actual)

PRIMARY OUTCOMES:
The Stroke Rehabilitation Assessment of Movement Measure (STREAM) | Patients were evaluated immediately before rehabilitation, and immediately after rehabilitation service, which lasted 4-10 days on average.
  The Stroke Rehabilitation Assessment of Movement Measure (STREAM) is a scale with scores ranging from 0 to 70, which is used to provide an understanding of the levels of movement and quality of hemiplegic patients.

SECONDARY OUTCOMES:
The Functional Independent Measurement (FIM) | Patients were evaluated immediately before rehabilitation, and immediately after rehabilitation service, which lasted 4-10 days on average.
  The Functional Independent Measurement (FIM) is 18-item scale and is scored from 18 (total assistance in all areas) to 126 (complete independence). FIM consists of 13 motor (or physical) and 5 social-cognitive items, assessing self care, sphincter control, transfer, locomotion, communication, social interaction, and cognition. The results from the first 13 items (FIM motor) are summed to develop a motor score with a range of 13 to 91, and these items were used in this study.
Mini-Mental State Examination (MMSE) | Patients were evaluated immediately before rehabilitation, and immediately after rehabilitation service, which lasted 4-10 days on average.
  Mini-Mental State Examination (MMSE) is a scale with scores ranging from 0 to 30, which allows the cognitive levels to be determined by examining the patient's orientation, recording memory, attention and calculation, recall, and language parameters. The score of 0 indicates that the patient has no cognitive functions, and the score of 30 indicates that the patient has a high level of cognitive functions.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided